CLINICAL TRIAL: NCT01567735
Title: An Open-Label, Single-Arm Phase III Study to Evaluate the Efficacy, Safety and Tolerability of TMC435 in Combination With PegIFN Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment-Naïve or Treatment-Experienced, Chronic Hepatitis C Virus Genotype-4 Infected Subjects
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of TMC435 in Combination With PegIFN Alfa-2a (Pegasys) and Ribavirin (Copegus) in Treatment-Naïve or Treatment-Experienced, Chronic Hepatitis C Virus Genotype-4 Infected Patients
Acronym: RESTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100695; TMC435HPC3011 (Other: Janssen R&D Ireland); 2011-004097-29 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-03-30 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435HPC3011; TMC435
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- TMC435 (Experimental)
  Interventions: Drug: TMC435

INTERVENTIONS:
Drug: TMC435 — Type=exact number, unit=mg, number=150, form=capsule, route=oral use. TMC435 capsule is taken once daily for 12 weeks.

SUMMARY:
The purpose of this study to evaluate the efficacy, safety and tolerability of TMC435 in combination with Peginterferon alfa-2a (PegINF alfa-2a) and ribavirin (RBV) in both treatment-naïve and treatment experienced, chronic hepatitis C (HCV) virus, genotype-4 infected patients.

DETAILED DESCRIPTION:
This is an open-label (both participant and investigator know the name of the medication given at a certain moment), single arm Phase III study, with 3 subpopulations: treatment naive, previous HCV relapser and previous HCV non-responders. The study will consist of 3 phases: a screening phase of maximum 6 Weeks, an open-label treatment phase of 24 to 48 Weeks for treatment naive patients and relapsers (response guided treatment) and 48 Weeks for non-responders, followed by a 24 Week follow-up period. The duration of participation in the study for an individual participant will be up to 54 to 78 (including screening).

Part Ia: All participants will receive 12 Weeks of triple therapy with TMC435 (150mg once daily [q.d.]), PegINF-alfa-2a (180µg per Week) and RBV (1000 to 1200 mg per day, based on weight), followed by 12 Weeks of PegINF-alfa-2a (180µg per Week) and RBV (1000 to 1200 mg per day, based on weight).

Part Ib: Participants who will need to continue treatment for another 24 Weeks (non-responders + treatment naive and relapser patients who need to continue treatment according to the response guided treatment criteria) will receive an additional 24 Weeks of PegINF-alfa 2a (180 mg per Week) and RBV (1000 to 1200 mg per day, based on weight).

Part II: 24 Week follow-up period for all participants, starting after Week 24 or Week 48.

In Part Ia, participants will have to come for 6 visits during the first month, followed by a visit once every month until Week 24 (in total 11 visits- Day1, day 3, Day 7, Day 14, day 28, Week 8, Week 12, Week 16, Week 20 and Week 24) at which safety, efficacy and tolerability will be checked.

In Part Ib, participants will have to come for 4 additional visits (Week 28, Week 36, Week 42 and Week 48) at which safety, tolerability and efficacy will be checked In the follow-up period, participants will have to come for an additional 3 visits (either Week 28, Week 36 and Week 28 or Week 52, Week 60 and Week 72) at which safety and efficacy will be checked.

Participants who withdraw prematurely will have a visit at withdrawal, 4 Weeks after withdrawal and then every 12 Weeks until 72 Weeks after baseline at which safety will be checked.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 4 Hepatitis C virus (HCV) infection (confirmed at screening)
* Plasma HCV ribonucleic acid (RNA) of >10,000 IU/mL at screening
* Participants should be either treatment-naïve or treatment-experienced (non-responder or relapser) with adequate documentation of previous response
* Participants must have voluntarily signed an Informed Consent Form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study. To participate in the optional pharmacogenomic component in this study (exploratory host genotyping), participants must have voluntarily signed a separate ICF for this component (where local regulations permit). Refusal to give consent for this component does not exclude a participant from participation in the core study.
* Participants must have had a liver biopsy within 3 years prior to screening (or between screening and baseline visit) with histology consistent with chronic HCV infection

Exclusion Criteria:

* Has an infection/co-infection with non-genotype 4 HCV
* Has a co-infection with Human Immunodeficiency Virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibodies test at screening).
* Has any of the following laboratory abnormalities:

  1. Platelet count <90,000/mm3;
  2. Absolute neutrophil count (ANC) <1500 cells/mm3 (Blacks: <1200 cells/mm3);
  3. Hemoglobin <12 g/dL for women and <13 g/dL for men;
  4. Creatinine >1.5 mg/dL;
  5. ALT and/or AST >10 x upper limit of normal (ULN);
  6. Total serum bilirubin >1.5 x ULN;
  7. Alpha-fetoprotein [AFP] >50 ng/mL;
  8. Albumin plasma concentration <3.5 g/dL;
  9. Prothrombin time (PT) expressed as international normalized ratio (INR) >1.5. Note: retesting of abnormal laboratory values that leads to exclusion will be allowed once using an unscheduled visit during the screening period to assess eligibility.
* Used disallowed concomitant therapy
* Has evidence of hepatic decompensation (history or current evidence of ascites, bleeding varices or hepatic encephalopathy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2014-03-20 (Actual); Study Completion 2014-03-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving sustained virologic response 12 weeks after planned end of treatment (SVR12) | Up to Week 60
  The primary objective is to evaluate the efficacy of TMC435 in combination with pegylated interferon alpha-2a (PegIFNα 2a)/ribavirin (RBV) with respect to the proportion of participants with chronic HCV-4 infection achieving SVR 12 weeks after planned end of treatment (SVR12) in the overall population as well as in the different subpopulations (treatment-naïve, previous relapsers and previous non-responders).

SECONDARY OUTCOMES:
Efficacy of TMC435 with respect to proportion of participants achieving sustained virologic response 24 weeks after planned end of treatment (SVR24) | Up to Week 72
  To evaluate the proportion of participants with SVR24, assessed 24 weeks after the planned end of treatment, in the overall population as well as in the different subpopulations
On-treatment virologic response | Week 4, Week 12, Week 24, Week 36, Week 48
  To evaluate on-treatment virologic response at all time points with focus on Week 4, Week 12, Week 24, Week 36, Week 48, in the overall population as well as in the different subpopulations.
On-treatment virologic failure | Up to Week 48
  To evaluate on-treatment virologic failure in the overall population as well as in the different subpopulations.
Evaluation of the viral breakthrough rate | Up to Week 48
  To evaluate the viral breakthrough rate on TMC435 in combination with PegIFNα-2a/RBV in the overall population as well as in the different subpopulations
Evaluation of viral relapse rate | Up to Week 48
  To evaluate the relapse rate after TMC435 in combination with PegIFNα-2a/RBV in the overall population as well as in the different subpopulations
Evaluation the safety and tolerability | Up to Week 72
  To evaluate the safety (includes adverse events, clinical lab tests, ECG and vital signs) and tolerability of TMC435 in combination with PegIFNα-2a/RBV

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (8):
- Belgium (3):
  - Antwerp
  - Brussels
  - Edegem
- France (5):
  - Clichy
  - Créteil
  - Lyon
  - Paris
  - Villejuif

REFERENCES:
- [Result] Moreno C, Hezode C, Marcellin P, Bourgeois S, Francque S, Samuel D, Zoulim F, Grange JD, Shukla U, Lenz O, Ouwerkerk-Mahadevan S, Fevery B, Peeters M, Beumont M, Jessner W. Efficacy and safety of simeprevir with PegIFN/ribavirin in naive or experienced patients infected with chronic HCV genotype 4. J Hepatol. 2015 May;62(5):1047-55. doi: 10.1016/j.jhep.2014.12.031. Epub 2015 Jan 14. PMID 25596313